CLINICAL TRIAL: NCT04718701
Title: Anlotinib Plus Toripalimab and Nab-paclitaxel in Patients With Locally Advanced or Metastatic Pancreatic Cancer: an Open-label, Non-randomized, Phase Ⅱ Study
Brief Title: Anlotinib, Toripalimab and Nab-paclitaxel in Locally Advanced/Metastatic Pancreatic Cancer
Acronym: ATNPA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-SR-496
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Neoplasm; Metastatic Pancreatic Cancer; Locally Advanced Pancreatic Adenocarcinoma
Keywords: Locally advanced pancreatic cancer; Metastatic pancreatic cancer; Anlotinib; Toripalimab; Nab-paclitaxel; Chemotherapy; PD-1 blockade; multi-targeted TKI
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Patients who failed first-line therapy with locally advanced or metastatic pancreatic cancer will be assigned to receive anlotinib plus toripalimab and nab-paclitaxel as second-line or maintenance treatment.
  Interventions: Drug: Anlotinib+Toripalimab+Nab-paclitaxel

INTERVENTIONS:
Drug: Anlotinib+Toripalimab+Nab-paclitaxel — Using combination treatment of anlotinib (12 mg, po. qd.) plus toripalimab (240 mg, ivgtt. q3w.) and nab-paclitaxel (260 mg/m2, ivgtt, q3w) with every 3 weeks as a cycle.
  Other Names: combination therapy

SUMMARY:
This is an open-label, non-randomized, single-arm phase Ⅱ study aiming to evaluate the efficacy and safety profile of above-mentioned combination strategy in first-line therapy-failed advanced pancreatic cancer. Totally 53 patients with locally advanced or metastatic pancreatic cancer are to be enrolled and receive anlotinib plus toripalimab and nab-paclitaxel.

DETAILED DESCRIPTION:
Anlotinib Hydrochloride Capsules (12 mg orally, once daily before breakfast; CTTQ, Lianyungang, Jiangsu, China), Toripalimab (240 mg intravenously, once every 3 weeks; Shanghai Junshi Biosciences Co., Ltd., Shanghai, China) and Nab-paclitaxel (125 mg/m2 intravenously, twice every 3 weeks; CSPC, Shijiazhuang, Hebei, China) are to be administered as a second-line therapy at most 6 cycles. Patients assessing as CR/PR/SD continue to receive a maintenance treatment including anlotinib and toripalimab until disease progression, intolerable toxicity, patient request for discontinuation for up to two years.

Observations and assessments will be conducted before treatment, on day 7, 21 of cycle 1, on day 21 of cycle 2, every 2 cycles (42 days) during following cycles and after treatment. Follow-up for survival status and subsequent antineoplastic therapy data collecting will be performed by telephone interview or face-to-face every 6 weeks after treatment until disease progression, death or end of the study (whichever occurs first).

Using 2.9 months served as a control, the expected median PFS of patients treated with anlotinib plus toripalimab and nab-paclitaxel in this study is prespecified as 4.5 months. Significance level α=0.05 (two-tailed) and test power (1-β)=0.80 are used for sample size calculation by PASS (Power Analysis and Sample Size) software. Taking a 20% drop-out rate into consideration, the sample size is approximately 53 patients. An interim analysis will be performed using a Lan-DeMets Pocock type boundary to assess the futility and efficacy when approximately half of the predetermined sample size is allocated. If the interim analysis results indicate that the study is of futility and the benefit/risk ratio is significantly worse, the trial will be terminated by the investigators. Otherwise, the trial will continue until the full sample size of 53 has been accumulated.

Efficacy is to be analyzed in the full analysis set (FAS), the response evaluable set (RES) and per-protocol set (PPS). Safety is to be analyzed in safety set (SS) including all assigned patients who receive at least one dose of study combined therapy and have safety records of medication. Statistical descriptions of subject distribution, demographic data and baseline characteristics will be performed. For study endpoints, the Kaplan-Meier method is to be applied for the PFS and OS curve with estimation for median PFS, median OS and 95% CI. ORR= (CR+PR) / sample size×100%; DCR= (CR+PR+SD) / sample size×100%. The 95% CI of the ORR and DCR are to be calculated by exact binomial method based on the F distribution. ECOG PS scores and QoL scores will be described at each visit time. For safety analysis, only treatment emergent adverse event (TEAE) will be included and analyzed in this experiment, which is defined as AEs that are post-dose or heavier than the baseline. Medical Dictionary for Regulatory Activities (MedDRA), system organ class (SOC), preferred terms (PT) and NCI CTCAE 5.0 will be used to standardize and classify all adverse events and summarize the incidence of AEs and association with treatments. Vital signs, ECG, and laboratory evaluation results will be compared and analyzed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-75.
2. Locally advanced / metastatic pancreatic cancer confirmed by histopathology.
3. Life expectancy ≥ 3 months.
4. Treatment failure after first-line monotherapy or combination chemotherapy (at least one cycle) or after adjuvant / neoadjuvant therapy.
5. At least one measurable tumor lesions without local treatment such as radiotherapy according to the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1); or tumor lesions in target area of previous radiotherapy confirmed progress.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
7. Adequate organ and bone marrow function.
8. Female of childbearing age must have a negative pregnancy test (serum or urine) within 7 days prior to enrolment. Males and females voluntarily use appropriate methods of contraception during study.
9. Voluntary provision of informed consents.

Exclusion Criteria:

1. Previous treatment with anlotinib, toripalimab or nab-paclitaxel.
2. Coexistence with intestinal perforation, massive intestinal gas, acute intestinal obstruction, severe infection and so on.
3. Multiple factors affecting oral medication such as inability to swallow, chronic diarrhea and intestinal obstruction.
4. Active bleeding of primary lesions within 2 months.
5. History of congenital/acquired immunodeficiency or organ transplantation.
6. Symptomatic brain metastases or meningeal metastases.
7. Existence with anyone of the following conditions: severe cardiovascular diseases, liver diseases, psychiatric disorders, poorly-controlled diabetes (fasting blood glucose>10mmol/L) or hypertension (systolic blood pressure≥150 mmHg and/ or diastolic blood pressure≥100 mmHg), active or uncontrolled severe infections, significant bleeding tendencies or under thrombolytic or anticoagulant treatment; occurrence of arterial and venous thrombotic events or clinically significant cardiovascular events within 6 months before enrollment；routine urinalysis showing urine protein ≥ ++ and confirmed 24-hour urine protein quantification > 1.0 g.
8. Known to be allergic to the test drug.
9. Pregnant or breastfeeding female patients
10. Other serious hazards to the safety of patients or complications that affect the study according to the judgment of the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months.
  From allocation to first disease progression confirmed by imaging modalities or all cause death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months.
  From allocation to any cause death or last follow-up.
Object response rate (ORR) | Up to 24 moths.
  Containing the incidence of complete response (CR) and partial response (PR).
Disease control rate (DCR) | Up to 24 months.
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD).
Quality of life (QoL) | up to 24 months.
  QoL refers to EORTC QLQ-C30 (version 3, Chinese version), and will be recorded in case report form (CRF) by observing clinical symptoms and scoring related examination before and after study treatment.
The incidence and severity of adverse events (AEs) and severe adverse events (SAEs) | Up to 24 months.
  AEs and SAEs will be graded and recorded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC, version 4.0). AEs are defined as any adverse medical events that occur in subjects from initiation of allocation up to 30 days after the last administration. SAEs are defined as all adverse medical events at any drug dose that result in a fatal, life-threatening event or prolonged hospital stay, permanent disability or other important medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xiang Liu, Physician, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD and all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication.
Access Criteria: IPD will be shared to other related clinical trials or systematic review after reviewing requests by chief investigator and examiners.